CLINICAL TRIAL: NCT02947802
Title: Sugar Sweetened Beverage Labeling Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Responsible Party: Principal Investigator, Leslie John, Principal Investigator, Harvard University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB16-1585
Record Dates: First submitted 2016-10-26; First posted 2016-10-28 (Estimated); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Consumer Behavior
MeSH Terms: conditions — Consumer Behavior

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Consumer Support (Experimental): Participants will be presented with three labels: a calorie label, a textual warning label and a textual warning label with corresponding graphic images and will be asked to rate their support for each label on a 1 (not at all) to 7 (a great deal) scale.
  Interventions: Other: Control condition
- Consumer Support with Effectiveness Info (Experimental): Participants will be presented with three labels: a calorie label, a textual warning label and a textual warning label with corresponding graphic images and will be asked to rate their support for each label on a 1 (not at all) to 7 (a great deal) scale. Participants will also receive effectiveness information- how each label influenced the purchasing of sugar sweetened beverages- from a recent field experiment.
  Interventions: Other: Effectiveness of Labels in Reducing Purchasing of Sugar Sweetened Beverages

INTERVENTIONS:
Other: Effectiveness of Labels in Reducing Purchasing of Sugar Sweetened Beverages — In one of our parallel assigned conditions participants will receive additional information (e.g., an intervention) of effectiveness information. These consumers will learn how effective these labels were in reducing the purchasing of sugar sweetened beverages in a recent study.
  Arms: Consumer Support with Effectiveness Info
Other: Control condition — In one of our parallel assigned conditions participants will receive no additional information and be asked to rate their support for the label.
  Arms: Consumer Support

SUMMARY:
This is an online survey assessing consumer support for different labeling policies related to sugar sweetened beverages. The investigators will present consumers with three labels that are being considered for sugar sweetened beverages: a calorie label, a text warning label that says "Warning drinking beverages with added sugar(s) can lead to health problems like obesity, diabetes and tooth decay" and a graphic warning label that includes graphic images to correspond with each of the health problems listed with the text warning. The investigators will ask participants their support for each label. The investigators will also see if support for the labels change after learning of the effectiveness of these labels. The investigators will share the results of a recent field study that suggested calorie and textual warning labels had no influence on the purchasing of sugar sweetened beverages while the graphic label decreased purchasing by 11 percent.

ELIGIBILITY:
Inclusion Criteria:

* The investigators will recruit a nationally representative sample using ClearVoice, a company that recruits online survey takers.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2016-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Rate Support of a Label on a 1 (not at all) to 7 (a great deal) Scale. | Immediately following the presentation of the labels.
  Participants will rate their support of the label on a 1 (not at all) to 7 (a great deal)

CONTACTS AND LOCATIONS:
Locations (1):
- Harvard University, Cambridge, Massachusetts, United States

REFERENCES:
- [Derived] Donnelly GE, Zatz LY, Svirsky D, John LK. The Effect of Graphic Warnings on Sugary-Drink Purchasing. Psychol Sci. 2018 Aug;29(8):1321-1333. doi: 10.1177/0956797618766361. Epub 2018 Jun 18. PMID 29912624
- Available data/document: Study Instrument (Online Survey) — https://hbs.qualtrics.com/SE/?SID=SV_1LdkKR5P4DyCevH — This is the online survey participants will complete.